CLINICAL TRIAL: NCT02693795
Title: Baduanjin Exercise Prevents Post-Myocardial Infarction Left Ventricular Remodeling (BE-PREMIER Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, shuai Mao, Director, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BE-PREMIER trial
Record Dates: First submitted 2016-02-14; First posted 2016-02-29 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; left ventricular remodeling
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baduanjin exercise group (Experimental): The participants randomized to Baduanjin exercise will collectively practice at cardiac rehabilitation centre in Guangdong Provincial Hospital of Chinese Medicine. A detailed description of a standardized Baduanjin exercise protocol complied with the "Health Qigong Baduanjin Standard" enacted by the General Administration of Sports in 2003. Each Baduanjin exercise session lasts 45 minutes and continues twice per week for 12 weeks.
  Interventions: Other: Baduanjin exercise
- usual exercise control group (Active Comparator): Participants allocated to the usual exercise control group receive a closely supervised, group-format aerobic exercise program located on cardiac rehabilitation centre lasting 3 month. The program is consistent with the current recommended guidelines of moderate intensity exercises for MI.
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: Baduanjin exercise — A detailed description of a standardized Baduanjin exercise protocol complied with the "Health Qigong Baduanjin Standard" enacted by the General Administration of Sports in 2003.
  Arms: Baduanjin exercise group
Other: aerobic exercise — Participants allocated to the usual exercise control group receive a closely supervised, group-format aerobic exercise program located on cardiac rehabilitation centre lasting 3 month. The program is consistent with the current recommended guidelines of moderate intensity exercises for MI.
  Arms: usual exercise control group

SUMMARY:
Left ventricular (LV) remodeling following myocardial infarction (MI) is an established prognostic factor for adverse cardiovascular events and the leading cause of heart failure. Empirical observations suggests that Baduanjin exercise, an important component of traditional Chinese Qigong, exert potential impacts on cardiopulmonary function. However, the impact of a Baduanjin exercise-based cardiac rehabilitation program for patients recovering from recent MI has yet to be assessed. The aim of this trail is to evaluate whether Baduanjin exercise would prevent the maladaptive progression to adverse LV remodeling in patients following MI.

DETAILED DESCRIPTION:
The increasing evidence indicates that exercise after a MI is associated with decreases in LV end-diastolic/ systolic volumes and increases in LV ejection fraction (LVEF), improvement in activity tolerance and quality of life, and reduction in the overall and cardiovascular-related mortality. However, on account of the heterogeneity in exercise intervention, limitation in methodology, and the varied characteristics of study populations, some other trials reported that post-MI exercise does not alter LV remodeling or cardiac function. Thus, more strict randomized controlled studies are needed to evaluate the benefits of exercise after MI and provide more indisputable evidence for guidelines and health professionals.

As an important component of Chinese Qigong exercises, Baduanjin exercise has origins in ancient martial arts that have been practiced for thousands of years. It is a combination of moderate-intensity physical activity, meditation, and body awareness, which designed to improve holistic health. Baduanjin exercise can systematically exert the movable joints and muscle, enhance cardiopulmonary functions, and concurrently modulate mind and spirit, ultimately achieve the integration of mind and body. Many clinical studies have demonstrated the beneficial effects of Baduanjin exercise on decreasing cholesterol and triglyceride concentrations, controlling systemic hypertension, stabilizing glucose and glycosylated hemoglobin levels. Some review articles have described Baduanjin exercise as a therapy with potential to exert positive impacts on cardiopulmonary function. Additionally, several recent studies have proven the benefits of Baduanjin exercise including preventing ischemic stroke, relieving pain and stiffness, and improving sleep quality and psychological well-being. However, it is not known if Baduanjin exercise could be a feasible approach for post-MI individuals because the scientific basis for this intervention is limited. To address a research gap, the BE-PREMIER (Baduanjin Exercise PREvents post-Myocardial Infarction left vEntricular Remodeling) trial is designed and to assess LV remodeling in clinically stable post-MI patients after a 12-week period of Baduanjin exercise-based cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of MI who has successful revascularization after the symptom onset;
2. Aged 18 years or over and under 80 years;
3. Availability to attend sessions twice a week over a 12-week period;
4. Physical aptitude to participate in a Baduanjin exercise -based cardiac rehabilitation program.

Exclusion Criteria:

1. Inability or difficulty to exercise
2. Prior history of practicing Qigong (Taiji or Baduanjin exercise, etc);
3. Presence of unstable angina, detectable myocardial ischemia (at rest or on exertion), significant valvular disease, and hypertrophic cardiomyopathy;
4. Severe symptomatic congestive heart failure (NYHA cardiac function class IV or left ventricular ejection fraction≤35%);
5. Severe pulmonary disease, musculoskeletal system diseases, other comorbidities precluding physical activity;
6. Life-threatening diseases with limited life expectancy <1 year;
7. Pregnant and lactating women;
8. Participation in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the percentage change from baseline to 6 months (%Δ) in echocardiographic LV end-diastolic volume index (LVEDVi) | baseline and 6 months
  the percentage change end-diastolic volume index (%)

SECONDARY OUTCOMES:
the change in echocardiographic measures of ventricular volumes (LV end-systolic/ diastolic volume) | baseline and 6 months
  LV end-systolic/ diastolic volume (mL)
The occurrence and composite of major adverse cardiac events (MACE) | baseline and 6 months
  defined as cardiogenic death, stroke, recurrent myocardial infarction, readmission on account of deterioration of congestive heart failure or unstable angina, target vessel revascularization
MacNew heart disease health-related quality of life questionnaire | baseline and 6 months
  in Units on a Scale
The short form 36 questionnaire | baseline and 6 months
  in Units on a Scale
The 6-minute walk test | from 3 to 6 months
  A 6-minute walk test measures the distance patients can quickly walk in 6 minutes. (in meters)
cardiopulmonary exercise test | from 3 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Minzhou zhang, M.D., Study Chair — 2nd Affiliated Hospital of Guangzhou University of Chinese Medicine

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chen MG, Liang X, Kong L, Wang J, Wang F, Hu X, He J, Zeng RX, Mao S, Guo L, Zhang MZ, Zhang X. Effect of Baduanjin Sequential Therapy on the Quality of Life and Cardiac Function in Patients with AMI After PCI: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2020 Jul 4;2020:8171549. doi: 10.1155/2020/8171549. eCollection 2020. PMID 32714423
- [Derived] Mao S, Zhang X, Shao B, Hu X, Hu Y, Li W, Guo L, Zhang M. Baduanjin Exercise Prevents post-Myocardial Infarction Left Ventricular Remodeling (BE-PREMIER trial): Design and Rationale of a Pragmatic Randomized Controlled Trial. Cardiovasc Drugs Ther. 2016 Jun;30(3):315-22. doi: 10.1007/s10557-016-6660-7. PMID 27106833